CLINICAL TRIAL: NCT05534217
Title: A Prospective, Randomized, Double-blind, Controlled Clinical Study of Corneal Debridement to Treat the Traumatic Corneal Abrasion
Brief Title: The Debridement To Treat The Traumatic Corneal Abrasion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022KYPJ139
Record Dates: First submitted 2022-08-05; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Corneal Abrasion
MeSH Terms: conditions — Corneal Injuries

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with traumatic corneal epithelial abrasions are treated by complete debridement of the corneal epithelium
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants didn't know where they were grouped,and the experimenters did not know about the trial either.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- debridement+traditional treatment (Experimental): The experimental group receives debridement of the abrasion wound before receiving traditional treatment including evofloxacin eye drops + befushu QID * for 14 days, four times a day, and the corneal contact lens was worn for 2 weeks.
  Interventions: Biological: corneal debridement of corneal abrasion
- traditional treatment (Active Comparator): The traditional group receives evofloxacin eye drops + befushu QID * for 14 days, four times a day, and the corneal contact lens was worn for 2 weeks.
  Interventions: Biological: corneal debridement of corneal abrasion

INTERVENTIONS:
Biological: corneal debridement of corneal abrasion — Surgical debridement for traumatic corneal epithelial abrasions

SUMMARY:
Patients who signed informed consent to participate in the study will receive corneal epithelial deplasia. The patient was instructed to follow up closely in the following year, and the recurrence of the patient was collected through wechat follow-up.

DETAILED DESCRIPTION:
Traumatic corneal abrasion (TCA) refers to the injury or defect of the corneal epithelium caused by a foreign object (such as a nail, a tree branch, etc.), which is characterized by severe eye pain accompanied by red eyes, blepharospasm, photophobia, tearing, and a distinct foreign body sensation. TCA is one of the common eye injuries and ophthalmic emergencies, accounting for about 5%-10% in ophthalmic emergencies. Methods: The investigators conducted a clinical trial in adult patients with corneal trauma at the Zhongshan Ophthalmology Center of Sun Yat-sen University. Patients who signed informed consent to participate in the study were provided with corneal epithelial debridement. Patients were instructed to follow closely for the following year, and a pain log of the patient was collected at the last ophthalmology clinic visit.

ELIGIBILITY:
Inclusion Criteria:

1. The affected eye is traumatic corneal epithelial abrasion, and the specific criteria are as follows: A: Damage caused by one of the three high risk causes of recurrent corneal epithelial exfoliation defined as fingernails, paper, or plant leaves; B: Monocular disease; C: Eye pain, tears, photophobia and foreign body sensation when injured; D: Local defect of corneal epithelium was found at the time of injury, and fluorescein sodium staining was positive; E: The time from injury to first diagnosis is less than 24 hours.
2. Be between the ages of 18 and 60.
3. Patients volunteered to participate in the study and signed the informed consent, showing good compliance.

Exclusion Criteria:

1. Corneal epithelial defect complicated with infection.
2. Patients with other ocular surface diseases (such as eyelid insufficiency, eyelid gland dysfunction, Sjogren's syndrome, bullae keratopathy, corneal dystrophy, drug induced corneal toxicity, etc.).
3. Pre-existing corneal disease (corneal degenerative disease or viral keratitis, etc.) or history of corneal surgery;
4. Long-term contact lens wearers.
5. Pregnant or lactating women; Severe impairment of heart, liver and kidney function; One who is mentally abnormal; People with other inflammatory or autoimmune diseases. Corneal epithelial defect complicated with infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 156 (Estimated)
Dates: Start 2022-12-31 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
wound recurrence | month 12 after treatment
  Wound recurrence during 12 months after treatment.

SECONDARY OUTCOMES:
Incidence of wound infection | week 1, week 2, month 1, month 2, month 3, month 6, month 9, and month 12.
  The incidence of wound infection during 12 months after treatment.
The grading of pain for eyes | week 1, week 2, month 1, month 2, month 3, month 6, month 9, and month 12.
  The degree of pain is evaluated during 12months after wounded. VRS（verbal rating scale）is used to evaluate the grading of pain,which is a line to describe the degrees of the pain that patients suffer from the disease, and the high scores is a worse outcome.
  The 5-point Verbal Rating Scale (VRS-5). （ ）Mild （ ）Discomforting （ ）Distressing （ ）Horrible （ ）Lxcruciaring
Corneal scar | week 1, week 2, month 1, month 2, month 3, month 6, month 9, and month 12.
  It is evaluated by the doctor in follow-up during 12 months. The haze of the corneal scar，and the high scores is a worse outcome.
  The degrees :
  0-clear cornea 0.5 - trace/just perceptible
  1. - easily seen with slit-lamp
  2. - moderate haze
  3. - pronounced haze, iris details still visible
  4. - "scarring", iris detail obscured (visible with pen torch)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhaohui Yuan, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No